CLINICAL TRIAL: NCT00620438
Title: Pharmacokinetic Interaction Between Coartem® and Either Nevirapine, Efavirenz or Rifampicin in HIV Positive Ugandan Patients
Brief Title: Drug Interaction Between Coartem® and Nevirapine, Efavirenz or Rifampicin in HIV Positive Ugandan Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Makerere University (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Concepta Merry, Infectious Diseases Institute, Makerere University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CPR 005
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Lumefantrine; Efavirenz; Nevirapine; Rifampicin; HIV
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Artemether, Lumefantrine Drug Combination; Nevirapine; stavudine, lamivudine, nevirapine drug combination; efavirenz; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): nevirapine arm
  Interventions: Drug: Lumefantrine-artemether and nevirapine
- 2 (Experimental): efavirenz arm
  Interventions: Drug: lumefantrine-artemether and efavirenz
- 3 (Experimental): Rifampicin arm
  Interventions: Drug: Lumefantrine-artemether and rifampicin

INTERVENTIONS:
Drug: Lumefantrine-artemether and nevirapine — Administration of lumefantrine 480mg co-formulated with artemether 80mg twice daily for three days to HIV positive patients receiving nevirapine 200mg twice daily as part of their antiretroviral treatment
  Other Names: Coartem; Triomune
  Arms: 1
Drug: lumefantrine-artemether and efavirenz — Administration of lumefantrine 480mg co-formulated with artemether 80mg twice daily for three days to HIV positive adults receiving efavirenz tablets 600mg once daily
  Other Names: Coartem; Sustiva
  Arms: 2
Drug: Lumefantrine-artemether and rifampicin — Administration of lumefantrine 480mg co-formulated with artemether 80mg twice daily for three days to patients receiving rifampicin as part of fixed dose combination therapy for tuberculosis
  Other Names: Coartem
  Arms: 3

SUMMARY:
There are increasing numbers of HIV-infected patients in sub-Saharan Africa receiving antiretroviral drugs and/or rifampicin based antituberculous therapy. HIV infected patients are at an increased risk of contracting malaria. Increasing resistance to anti-malarials such as chloroquine, amodiaquine, fansidar, sulphadoxine-pyrimethamine in East and West Africa has led the WHO to recommend artemether-lumefantrine (Coartem®- Novartis) as first line therapy for malaria for adults and children. As early as 2004, fourteen countries in sub-Saharan Africa had adopted this guideline as national policy.

There are no data on the interaction between Coartem® and any of the antiretroviral agents. Both components of Coartem® are substrates for the 3A4 isoform of cytochrome P450. Despite the lack of data, antiretroviral drugs and/or antituberculous drugs in addition to Coartem® are of necessity co-prescribed daily in the African setting. Nevirapine, efavirenz and rifampicin are known inducers of cytochrome P450 3A4. A technical consultation convened by WHO in June, 2004 concluded that additional research on interactions between antiretroviral and antimalarial drugs is urgently needed.

We propose to perform a suite of pharmacokinetic studies to evaluate these interactions in HIV infected Ugandan patients. The aim of these studies is to evaluate the pharmacokinetic interaction between Coartem® and commonly co-prescribed inducers of 3A4 i.e. nevirapine, efavirenz and rifampicin.

1. Comparison of steady state pharmacokinetics of Coartem® in HIV-infected patients prior to commencement of nevirapine and at nevirapine steady state
2. Comparison of steady state pharmacokinetics of Coartem® in HIV-infected patients prior to commencement of efavirenz and at efavirenz steady state
3. Comparison of steady state pharmacokinetics of Coartem® in Ugandan patients at rifampicin steady state and without rifampicin

DETAILED DESCRIPTION:
Coartem® is the combination of artemether and lumefantrine used for the treatment of uncomplicated falciparum malaria 1. This oral combination seems to be well-tolerated and is useful for treatment of multi-drug resistant Plasmodium falciparum. This unique anti-malarial agent combines the fast, but short-acting artemether with a less potent, but longer-acting lumefantrine. Original studies with the combination demonstrated safety and efficacy in adults and children with uncomplicated falciparum malaria. 2,3 Additional studies showed superiority with respect to parasite clearance time versus halofantrine,4 chloroquine5, and mefloquine6. Coartem® also demonstrated a faster reduction in parasite burden after 24-hours versus halofantrine4, chloroquine5 (in adults), chloroquine (in children) 7, and mefloquine6. Various other studies have shown artemether-lumefantrine to have a superior 28-day cure rate, as well as time to fever resolution compared to other antimalarial agents.1 Both components of Coartem® were discovered in China. Artemether was isolated from sweet wormwood, Atemisia annua, which has been used in traditional Chinese medicine for over 2000 years 1. Lumefantrine is a synthetic compound, which has structural and physiochemical characteristics; and a mode of action similar to other antimalarials, including quinine, mefloquine, and halofantrine 8. In vitro, the two antimalarial agents show synergistic activity against P.falciparum. Based on both in vitro and in vivo studies, a 1:6 ratio of artemether to lumefantrine has been described as optimal. Thus, the tablets are manufactured as 20mg artemether and 120mg lumefantrine. 8 Currently there are two recommended dosing regimen for adults and children above 35 kg; or 12 years of age or older. In partially immune patients, a 4-dose regimen is recommended. Four tablets as a single dose should be taken at time of diagnosis and then again at 8, 24, and 48 hours post-initial dose. A different regimen is recommended for either non-immune patients or patients in areas where multi-drug resistance to falciparum malaria is a problem. This is a 3-day regimen consisting of 4 tablets as a single dose given at the time of diagnosis, 8 hours later and then twice daily for the following two days. 1

Antimalarial Activity and Mechanism of Action: 1, 8 The antimalarial activity of artemether and that of its active metabolite, dihydroartemisinin (DHA) have been extensively studied in vitro. These are very potent antimalarial compounds. The IC50 of artemether ranges from 0.1 to 20 nmol/L and the IC50 for DHA ranges from 0.1 to 15 nmol/L. In vitro studies have shown artemether to be 2 to 3 times less active than its metabolite, DHA.

The exact mechanisms of action of artemether and lumefantrine are unknown, but both agents appear to act on the parasite's organelles. Artemether's action depends on its endoperoxide bridge, which interacts with heme iron to cause free radical damage to the malaria parasite. Lumefantrine most likely interferes with heme polymerization, which is a critical detoxifying pathway for the malaria parasite. Both agents may have secondary actions that include inhibition of parasite nucleic acid and protein synthesis; however, these actions have not been well-described.

The varied pharmacokinetic profiles of the two antimalarial agents appear to create a synergistic effect. Artemether works rapidly to decrease the parasite load and improve patients' clinical symptoms. Lumefantrine is long-acting and appears to prevent recrudescence (reappearance of the disease after inadequate or failed drug therapy). The different actions of the two agents may also reduce the emergence of resistance. Artemether and DHA have been shown to decrease parasite burden by about 104 per asexual life cycle in about 2 days. Thus, the 3-day course of the combination therapy can potentially decrease the parasite burden by about 108.

Drug Interactions Pharmacokinetic and electrocardiographic interactions between artemether-lumefantrine and the mefloquine were studied in 42 healthy volunteers. Like artemether-lumefantrine, mefloquine is a substrate for CYP 3A4; however, it is also a potential CYP 3A4 inhibitor. Pharmacokinetic parameters for artemether, DHA, and mefloquine were unchanged; however, lumefantrine concentrations decreased by 30-40% when given with mefloquine. The clinical significance of this interaction is not known. Co-administration of the antimalarial agents resulted in no increased adverse effects. 13

An additional study evaluated the effects of concomitant administration with ketoconazole, a potent CYP 3A4 inhibitor, and artemether-lumefantrine. The study was carried out in 16 healthy volunteers who received single doses of artemether-lumefantrine either alone or in combination with multiple doses of ketoconazole. Artemether, DHA, and lumefantrine pharmacokinetics were altered by ketoconazole. AUC and Cmax increased for all three compounds and terminal half-life increased for artemether and DHA. None of the changes in PK parameters were greater than those changes observed in healthy volunteers taking artemether-lumefantrine with a high fat meal (i.e. a 16-fold increase in AUC). There was no increase in observed side effects or electrocardiographic changes. Dosage adjustments do not appear to be necessary with concomitant ketoconazole administration.14

A study of 42 healthy Caucasian volunteers was conducted to investigate pharmacokinetic or electrocardiographic effects of concomitant administration of IV quinine and artemether-lumefantrine. QTc prolongation was not associated with artemether-lumefantrine administration alone; however transient increases in QTc interval were noted in the combination groups. PK variables for lumefantrine and quinine were unchanged, but artemether and DHA plasma concentrations decreased with concomitant quinine administration. The exact mechanism for this decrease could not be explained for the results of this study.15

Artemether is metabolized via CYP 3A4 to dihydroartemisinin (although both compounds have antimalarial activity, dihydroartemisinin has greater potency). Induction of CYP 3A4 would increase dihydroartemisinin but decrease artemether.

Study objectives General objective To evaluate the pharmacokinetic interaction between Coartem® and commonly co-prescribed inducers of 3A4 i.e. nevirapine, efavirenz and rifampicin in HIV positive patients.

Specific objectives

1. To compare the steady state pharmacokinetics of Coartem® in HIV-infected patients prior to commencement of nevirapine and at nevirapine steady state
2. To compare the steady state pharmacokinetics of Coartem® in HIV-infected patients prior to commencement of efavirenz and at efavirenz steady state
3. To compare the steady state pharmacokinetics of Coartem® in Ugandan patients at rifampicin steady state and without rifampicin therapy

ELIGIBILITY:
Inclusion Criteria:

* Age over eighteen years
* Ability to provide full written informed consent
* Confirmed diagnosis of HIV infection

Exclusion Criteria:

* Haemoglobin < 8g/dl
* Liver and renal function tests > 3 times the upper limit of normal
* Pregnancy
* Use of known inhibitors or inducers of cytochrome P450 or P-glycoprotein.
* Use of herbal medications (information will be obtained from patients' medication history through interview with the patient)
* Abnormal EKG ie QTc (Rate adjusted QT interval) >450ms (men) or >470ms (women)
* Intercurrent Illness including malaria
* Known hypersensitivity to artemisinin-derivatives, halofantrine or lumefantrine
* History of cardiac disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of lumefantrine in patients receiving either nevirapine, efavirenz or rifampicin | 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Concepta Merry, PhD, Principal Investigator — Trinity Colleg Dublin
Locations (1):
- Infectious Diseases Institute, Makerere University, Kampala, Uganda

REFERENCES:
- [Derived] Hoglund RM, Byakika-Kibwika P, Lamorde M, Merry C, Ashton M, Hanpithakpong W, Day NP, White NJ, Abelo A, Tarning J. Artemether-lumefantrine co-administration with antiretrovirals: population pharmacokinetics and dosing implications. Br J Clin Pharmacol. 2015 Apr;79(4):636-49. doi: 10.1111/bcp.12529. PMID 25297720